CLINICAL TRIAL: NCT04204564
Title: Vascular Implant Surveillance and Interventional Outcomes Network and the Vascular Quality Initiative Paclitaxel Safety Analysis
Brief Title: VISION and VQI Paclitaxel Safety Analysis
Acronym: VISION-VQI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Vermont Medical Center (Other)
Collaborators: The Medical Device Epidemiology Network (MDEpiNet) (Unknown); Society for Vascular Surgery Patient Safety Organization (Other)
Responsible Party: Principal Investigator, Daniel Bertges, MD, Associate Professor of Surgery and Medicine, University of Vermont Medical Center
Other Study IDs: 1
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: PAD
Keywords: paclitaxel; drug coated balloon; drug eluting stent; perihpheral vascular intervention; registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- paclitaxel coated balloon angioplasty: Procedures with paclitaxel coated balloon angioplasty of the superficial femoral-popliteal artery
  Interventions: Device: pactlitaxel PAD device
- plain balloon angioplasty: Procedures with plain balloon angioplasty of the superficial femoral-popliteal artery
- paclitaxel eluting stent: Procedures with paclitaxel eluting stenting of the superficial femoral-popliteal artery
  Interventions: Device: pactlitaxel PAD device
- bare metal stenting: Procedures with bare metal self expanding stenting of the superficial femoral-popliteal artery

INTERVENTIONS:
Device: pactlitaxel PAD device — Peripheral vascular intervention on femoral-popliteal occlusive disease with paclitaxel and non-paclitaxel devices.
  Other Names: Medtronic INPact Admiral; Bard Lutonix; Cook Zilver PTX stent
  Groups: paclitaxel coated balloon angioplasty; paclitaxel eluting stent

SUMMARY:
Objectives

1. The VQI-VISION Paclitaxel Device Safety Analysis seeks to assess the comparative safety of paclitaxel-coated balloons and stents in the treatment of PAD through analysis of the Vascular Quality Initiative (VQI) Peripheral Vascular Intervention (PVI) registry module with linkage to claims. By linking VQI patients to Medicare claims retrospectively from 2012 to 2016, we will be able to identify additional paclitaxel devices enabling longitudinal follow-up of mortality out to 5 years for paclitaxel-eluting stents and 3 years for paclitaxel-coated balloons.
2. To analyze factors associated with mortality, specifically comparing paclitaxel patients surviving vs. paclitaxel patients with mortality. The goal is to identify independent factors predictive of mortality in US pivotal trials and model registry data exposures with sufficient factors to track competing risk paradox and show emulation or not of mortality outcomes with both PTX and PTA exposures.
3. To confirm the effectiveness of paclitaxel devices by comparing reintervention for paclitaxel and non-paclitaxel devices. In-hospital mortality from open and percutaneous target vessel revascularization (TVR) will be reported to determine the impact of subsequent revascularizations on survival. Major amputation will be comparted for patients with chronic limb-threatening ischemia.

DETAILED DESCRIPTION:
The proposed safety analyses will evaluate two types of paclitaxel-coated interventional devices used to treat PAD and compare patient outcomes with propensity score-matched patients of similar risk who receive non-paclitaxel devices.

The primary outcome will be freedom from all-cause death using propensity-matched survival analysis.

Three principle analyses are planned:

1. Paclitaxel DCB (including the Bard Lutonix, Medtronic In.Pact Admiral, and Philips Spectranetics Stellarex DCB's) as compared with propensity-matched patients treated with plain balloons.
2. Paclitaxel delivering DES (Cook Zilver PTX) as compared with propensity-matched cases using bare-metal stents (BMS).
3. Patients treated with either Paclitaxel DCB or Paclitaxel DES compared with propensity-matched controls (with DCB patients matched to patients treated with plain balloons, and DES patients matched to patients treated with BMS).

Note that this analysis is planned at the device class level and is not intended to compare early or late mortality between specific devices or brands.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Date of index procedure is within 10/1/2012 to 12/31/2016
* Symptomatic disease ranging from intermittent claudication to chronic limb-threatening ischemia (including ischemic rest pain and/or tissue loss)
* Elective or urgent procedures

Exclusion Criteria:

* Aneurysmal disease of the superficial femoral or popliteal artery
* Treatment for acute limb ischemia
* Treatment of common femoral artery or profunda femoral artery occlusive disease
* Emergency procedures
* PVI and concomitant femoral endarterectomy, suprainguinal or infrainguinal bypass

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients, aged 65 or older, who underwent endovascular interventional treatment of the femoral or popliteal arteries for symptomatic PAD between 10/1/2012 and the latest available CMS dataset (12/31/2016) will be included.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2012-10-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
overall mortality | 1 year
  death from any cause
overall mortality | 3 years
  death from any cause
overall mortality | 5 years
  death from any cause

SECONDARY OUTCOMES:
target vessel revascularization (TVR) | 1-3-5 years
  repeat intervention on the SFA-popliteal artery including open or endovascular revascularization
Major amputation | 1-3-5 years
  Major amputation for patients with chronic limb-threatening ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bertges, MD, Principal Investigator — SVS VQI; Philip Goodney, MD, Study Director — SVS VQI; Art Sedrakyan, PhD, Study Director — Weill Medical College of Cornell University; Jens Jorgensen, Study Chair — SVS PSO

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Background] Columbo JA, Kang R, Hoel AW, Kang J, Leinweber KA, Tauber KS, Hila R, Ramkumar N, Sedrakyan A, Goodney PP. A comparison of reintervention rates after endovascular aneurysm repair between the Vascular Quality Initiative registry, Medicare claims, and chart review. J Vasc Surg. 2019 Jan;69(1):74-79.e6. doi: 10.1016/j.jvs.2018.03.423. Epub 2018 Jun 15. PMID 29914838
- [Background] Schillinger M, Minar E. Past, present and future of femoropopliteal stenting. J Endovasc Ther. 2009 Feb;16 Suppl 1:I147-52. doi: 10.1583/1545-1550-16.16.I-147. PMID 19317587
- [Background] Dick P, Wallner H, Sabeti S, Loewe C, Mlekusch W, Lammer J, Koppensteiner R, Minar E, Schillinger M. Balloon angioplasty versus stenting with nitinol stents in intermediate length superficial femoral artery lesions. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1090-5. doi: 10.1002/ccd.22128. PMID 19859954
- [Background] Chowdhury MM, McLain AD, Twine CP. Angioplasty versus bare metal stenting for superficial femoral artery lesions. Cochrane Database Syst Rev. 2014 Jun 24;2014(6):CD006767. doi: 10.1002/14651858.CD006767.pub3. PMID 24959692
- [Background] Eliason JL, Wainess RM, Proctor MC, Dimick JB, Cowan JA Jr, Upchurch GR Jr, Stanley JC, Henke PK. A national and single institutional experience in the contemporary treatment of acute lower extremity ischemia. Ann Surg. 2003 Sep;238(3):382-9; discussion 389-90. doi: 10.1097/01.sla.0000086663.49670.d1. PMID 14501504
- [Background] Earnshaw JJ, Whitman B, Foy C. National Audit of Thrombolysis for Acute Leg Ischemia (NATALI): clinical factors associated with early outcome. J Vasc Surg. 2004 May;39(5):1018-25. doi: 10.1016/j.jvs.2004.01.019. PMID 15111854
- [Background] Howard DP, Banerjee A, Fairhead JF, Hands L, Silver LE, Rothwell PM; Oxford Vascular Study. Population-Based Study of Incidence, Risk Factors, Outcome, and Prognosis of Ischemic Peripheral Arterial Events: Implications for Prevention. Circulation. 2015 Nov 10;132(19):1805-15. doi: 10.1161/CIRCULATIONAHA.115.016424. Epub 2015 Sep 8. PMID 26350058
- [Background] Baril DT, Ghosh K, Rosen AB. Trends in the incidence, treatment, and outcomes of acute lower extremity ischemia in the United States Medicare population. J Vasc Surg. 2014 Sep;60(3):669-77.e2. doi: 10.1016/j.jvs.2014.03.244. Epub 2014 Apr 24. PMID 24768362
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Mar 21;69(11):1465-1508. doi: 10.1016/j.jacc.2016.11.008. Epub 2016 Nov 13. No abstract available. PMID 27851991
- [Background] Oakes D, Feng C. Combining stratified and unstratified log-rank tests in paired survival data. Stat Med. 2010 Jul 20;29(16):1735-45. doi: 10.1002/sim.3921. PMID 20572124
- [Background] M Grambsch and TM Therneau, Proportional Hazards Tests and Diagnostics Based on Weighted Residuals, Biometrika 1994, 81(3): 515-526, https://doi.org/10.1093/biomet/81.3.515
- [Background] Royston P, Parmar MK. Restricted mean survival time: an alternative to the hazard ratio for the design and analysis of randomized trials with a time-to-event outcome. BMC Med Res Methodol. 2013 Dec 7;13:152. doi: 10.1186/1471-2288-13-152. PMID 24314264
- [Background] Parzen M, Lipsitz SR. A global goodness-of-fit statistic for Cox regression models. Biometrics. 1999 Jun;55(2):580-4. doi: 10.1111/j.0006-341x.1999.00580.x. PMID 11318217
- [Background] Heinze G, Wallisch C, Dunkler D. Variable selection - A review and recommendations for the practicing statistician. Biom J. 2018 May;60(3):431-449. doi: 10.1002/bimj.201700067. Epub 2018 Jan 2. PMID 29292533

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT04204564/SAP_000.pdf